CLINICAL TRIAL: NCT02515760
Title: Tumor-specific Effector T Cells in Non-small Cell Lung Cancer
Brief Title: Tumor-specific T Cells in Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other); Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. med. Seyer Safi, PD Dr. med. Seyer Safi, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S-515/2013
Record Dates: First submitted 2015-07-30; First posted 2015-08-05 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung cancer group (Experimental): Bone marrow puncture in patients with non-small cell lung cancer
  Interventions: Procedure: Bone marrow aspiration from the iliac crest; Device: Illinois bone marrow aspiration neddle
- Control group (healthy donors) (Experimental): Bone marrow puncture in healthy donors
  Interventions: Procedure: Bone marrow aspiration from the iliac crest; Device: Illinois bone marrow aspiration neddle

INTERVENTIONS:
Procedure: Bone marrow aspiration from the iliac crest
Device: Illinois bone marrow aspiration neddle

SUMMARY:
Non-small cell lung cancer is characterized by aggressive growth and treatment resistance. New approaches include immunotherapeutic strategies but spontaneous immune responses against tumor antigens remain unclear. The aim of this study is to characterize localization and frequencies of spontaneously induced memory T cells specific for a panel of tumor-associated antigens in peripheral blood and bone marrow of non-small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histology proven non-small cell lung cancer or a lesion suspicious of non-small cell lung cancer (lung cancer group)
* Healthy donors (control group)
* written informed consent

Exclusion Criteria:

* Autoimmune disease
* Patients receiving immunomodulatory drugs, e.g. tacrolimus
* Prior malignancy
* Pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-02; Primary Completion 2018-06 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Frequencies of tumor-specific T cells | 2 weeks postoperative
  % of all T cells

SECONDARY OUTCOMES:
Tumor-specific T cells location determined by Enzyme Linked Immuno Spot Assay (ELISPOT) analysis of peripheral blood and bone marrow samples from the same patient | 2 weeks postoperative
  location: peripheral versus bone marrow
Long-term survival | 5 years postoperative
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Seyer Safi, MD, PhD, Principal Investigator — Division Thoracic Surgery, Technical University of Munich, Munich, Germany
Locations (1):
- Division of Thoracic Surgery, Technical University of Munich, Munich, Germany, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamauchi Y, Safi S, Blattner C, Rathinasamy A, Umansky L, Juenger S, Warth A, Eichhorn M, Muley T, Herth FJF, Dienemann H, Platten M, Beckhove P, Utikal J, Hoffmann H, Umansky V. Circulating and Tumor Myeloid-derived Suppressor Cells in Resectable Non-Small Cell Lung Cancer. Am J Respir Crit Care Med. 2018 Sep 15;198(6):777-787. doi: 10.1164/rccm.201708-1707OC. PMID 29617574
- [Result] Safi S, Yamauchi Y, Hoffmann H, Weichert W, Jost PJ, Winter H, Muley T, Beckhove P. Circulating Interleukin-4 Is Associated with a Systemic T Cell Response against Tumor-Associated Antigens in Treatment-Naive Patients with Resectable Non-Small-Cell Lung Cancer. Cancers (Basel). 2020 Nov 24;12(12):3496. doi: 10.3390/cancers12123496. PMID 33255425
- [Result] Safi S, Yamauchi Y, Stamova S, Rathinasamy A, Op den Winkel J, Junger S, Bucur M, Umansky L, Warth A, Herpel E, Eichhorn M, Winter H, Hoffmann H, Beckhove P. Bone marrow expands the repertoire of functional T cells targeting tumor-associated antigens in patients with resectable non-small-cell lung cancer. Oncoimmunology. 2019 Oct 23;8(12):e1671762. doi: 10.1080/2162402X.2019.1671762. eCollection 2019. PMID 31741774
- [Result] Safi S, Yamauchi Y, Rathinasamy A, Stamova S, Eichhorn M, Warth A, Rauch G, Dienemann H, Hoffmann H, Beckhove P. Functional T cells targeting tumor-associated antigens are predictive for recurrence-free survival of patients with radically operated non-small cell lung cancer. Oncoimmunology. 2017 Sep 8;6(11):e1360458. doi: 10.1080/2162402X.2017.1360458. eCollection 2017. PMID 29147626